CLINICAL TRIAL: NCT04395729
Title: Functional Benefits of Multisite Surgery for the Upper Limb of Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Centre Médico-Chirurgical de Réadaptation des Massues Croix Rouge Française (Other)
Responsible Party: Sponsor
Other Study IDs: RETRO-CHIR
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy, Spastic; Cerebral Palsy, Dyskinetic; Infantile Hemiplegic Cerebral Palsy
Keywords: Upper limb; Contraction; Deformity; Multisite surgery; Treatment outcome
MeSH Terms: conditions — Cerebral Palsy; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to investigate the impact of individualized multisite neuro-orthopedic surgery of the upper limb in children with Cerebral Palsy on unilateral functional capacities and bimanual performance. The investigators also assessed the attainment of individualized goals and tracked any potential factors that may have an impact on final results.

DETAILED DESCRIPTION:
Cerebral Palsy is responsible for the most common neurological disorders in children. Although the primary lesion is non-evolutionary, the secondary consequences are evolutive, with neuro-orthopaedic degradation leading to soft tissue retraction and osteo-articular deformities. Hemiplegia occurs in approximately 30% of cases of Cerebral Palsy, and tone disorders (spasticity, dyskinesia) affecting the upper limb generally impact function, both in unilateral capacities (range of motion, dexterity, and fluidity of movement), and in bimanual performance. The focal treatment of spasticity by botulinum toxin injections, in combination with specific occupational therapy training, has proven to be effective in improving targeted functional goals. However, there is little evidence today of the effectiveness of treatment for the management of upper limb retraction and deformity, whether by stretching, orthosis/plaster or even surgery. And apart from its effectiveness on body structure, the functional effects of upper limb surgery in Cerebral Palsy have been little explored. The aim of the study is to investigate the impact of individualized multisite neuro-orthopedic surgery of the upper limb in children with Cerebral Palsy on unilateral functional capacities and bimanual performance, by using such tools as the Melbourne Assessment (Version 2) and the Assisting Hand Assessment (Version 5.0).

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years at time of surgical project
* Unilateral upper limb injury due to Cerebral Palsy
* Having undergone neuro-orthopaedic surgery of the upper limb with prior evaluation and comparative evaluation after surgery (6 months)

Exclusion Criteria:

- Refusal to process medical data concerning the child for research purposes

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (<18 years) with cerebral palsy, presenting with unilateral upper limb injury.
  Surgical procedures consisted of one and/or the other of the following interventions (possibility of combining several procedures depending on the highly individualized surgical decision): Adductor Pollicis Brevis Disinsertion, Flexor Carpi Ulnaris Disinsertion, Lengthening of fingers flexors, Transfer (FCU) to the Extensor Carpi Radialis Brevis, Pronator teres Disinsertion, Lengthening of elbow flexors, Wrist arthrodesis.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Melbourne Assessment - Version 2 | Available data up to 3 years before surgery and up to 2 years after surgery
  The Melbourne Assessment evaluates unilateral upper limb functional capacities for children between 2.5 and 15 years of age with neurological impairment.
  It takes into account movement patterns, by characterizing the articular positioning observed during movements, as well as the fluidity of movement. Through 14 items analyzed along 4 axes (range of motion, precision, dexterity and fluidity), this test explores unilateral capacities to reach, grasp, release and manipulate simple objects. The evaluation is filmed according to a standardized protocol analyzed on video. The scoring is based on the video and the result is expressed as 4 scores in % for the areas of: range of motion, precision, dexterity, fluidity of movement. The reliability of the tool proved to be very good for the total score, for intra-examiner reproducibility (R=0.97) and inter-examiner reproducibility as well (R=0.95).

SECONDARY OUTCOMES:
Assisting Hand Assessment - Version 5.0 | Available data up to 3 years before surgery and up to 2 years after surgery
  The Assisting Hand Assessment (AHA) evaluates the effectiveness of the use of the assistant hand in bimanual performance in children with unilateral impairment between 18 months and 18 years of age. The test is scored on the video recording of the bimanual performance observation session, through 20 items rated on a rating scale between 1=ineffective and 4=effective; the different AHA items characterize the general use of the upper limb, the use of the arm, the grasp-release domain, fine motor adjustment and coordination. The total raw score is reduced to an interval score between 0 and 100. The reliability of the AHA has been shown to be very good for the total score, both intra-examiner (CCI= 0.99) and inter-examiner (CCI= 0.98). A difference of 5 points on the interval scale 0-100 is considered a significant difference.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Chaléat-Valayer, MD, PhD, Principal Investigator — CMCR des Massues Croix rouge française
Locations (1):
- Croix rouge française Centre Médico-Chirurgical de Réadaptation des Massues, Lyon, France

IPD SHARING:
Plan to Share IPD: No